CLINICAL TRIAL: NCT03545399
Title: Essai Clinique randomisé en Double Aveugle Contre Placebo de l'évaluation de l'Effet d'un Extrait d'Algues Comestibles (Ulva Lactuca) Chez Des Volontaires Sains présentant Une anhédonie associée à Une Baisse de Moral
Brief Title: The Effect of an Edible Algal Extract (Ulva Lactuca) on the Component of Depression in Healthy Volunteers With Anhedonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CEN Biotech (Industry)
Collaborators: CEN Nutriment (Unknown); Biovet Conseil (Unknown); Amadeite SAS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1365
Record Dates: First submitted 2018-05-04; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Anhedonia in Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Single-centre double-blind randomized placebo-controlled clinical trial on parallel arms of two groups of 45 subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ulva Lactuca (Experimental): The subject is given a capsule containing a concentrated fraction of freeze-dried and crushed hydrosoluble extract of seaweeds. The dose tested of extract of seaweeds is of 6.45mg per kg weight. The daily dose is 3 capsules per day for subjects weighing between 50 and 70kg, 4 capsules per day for subjects weighing between 70 and 90kg and 5 capsules per day for subjects weighing between 90 and 110kg. The duration of the treatment is 12 weeks.
  Interventions: Dietary Supplement: Ulva Lactuca
- Placebo (Placebo Comparator): The subject is given a capsule looking alike that of the active product but containing no extract of seaweeds.The duration of the treatment is 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ulva Lactuca — The dose was taken with a glass of water during the evening meal once daily
  Arms: Ulva Lactuca
Dietary Supplement: Placebo — The dose was taken with a glass of water during the evening meal once daily
  Arms: Placebo

SUMMARY:
The effects of the seaweed extract were evaluated on the animal model equivalent of depression compared with a control group treated with the carrier (spring water) and a reference group treated with Imipramine and showed significative effect. This clinical trial was intended to confirm in humans the potential efficacy identified in animals. The primary objective was to compare against a placebo the effect of Ulva L.L extract in healthy volunteers whose anhedonia was characterized by a component of depression.

DETAILED DESCRIPTION:
The trial comprised three visits: a medical enrollment visit on D0, an intermediate visit on D28 and a final visit on D84. A psychologist made a telephone call after 7 days to check there was no sudden change in the subject's depressive state. During the visits, the subject was examined by a doctor and the psychometric tests were administered by a psychologist. Outside the visits, the subject was monitored by a self-reporting questionnaire in the manner described below.

After obtaining informed written consent and validating the inclusion and exclusion criteria, notably the absence of MDE as per DSM V, the investigator enrolled the subject in the trial. The physician described the subject's demographic and general clinical characteristics, the main medical and surgical history and any current treatment if those pathologies were still present, and any previous antidepressant, anxiolytic or neuroleptic treatments. The doctor asked the subject to complete the SHAPS and QIDS -SR questionnaires and item 7 of the HAM-D. The doctor then handed the subject self-evaluation questionnaires explaining how to complete them and the dates at which they were to be completed. The physician gave the patient a batch of the placebo or a batch of Ulva lactuca as per the randomization. The doctor told the subject a psychologist would be in touch after one week by telephone to check no DSM V severity criterion had arisen.

The investigating doctor saw the subject again at the four-week intermediate visit and at the final visit at the end of the 12th week of follow-up. The doctor collected the self-questionnaires at these visits and the same items as at the enrollment visit were recorded by the physician for describing how the items had evolved and notably the SHAP scale score, the QIDS-SR and item 7 of the HAM-D. In addition, the physician recorded the subject's satisfaction with the treatment evaluated on the PGII (Patient Global Improvement Impression), reported any undesirable affects and gave his/her own opinion on the efficacy of treatment using the Clinical Global Improvement Impression (CGII).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged between 18 and 65 years
* Presenting a anhedonia with a score ≥5 on the SHAPS Scale
* Declaring feeling low for at least 4 weeks characterised by a component of depression evaluated on the QIDS-SR
* Being able to apprehend and fill in the evaluation scales

Exclusion Criteria:

* Subject with a major depressive episode as per the DSM V scale, with a HAM D > 8, already on anxiolytic, antidepressor, neuroleptic or any other medicinal treatment liable to influence mood (e.g. benzodiazepines) in the last 30 days or using illegal psychotropic substances, or a with daily alcohol intake of more than three glasses of wine
* Presenting a psychiatric disorder or in state of post-traumatic stress or having had an electroconvulsive therapy in the last 6 months
* Female subject pregnant or breast-feeding or of childbearing age and not using effective means of contraception
* subject suffering from an allergy or intolerance to seafood products (fish, shellfish and seaweed)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Evolution of anhedonia in healthy subjects | 84 days
  The evolution of anhedonia in healthy subjects whose anhedonia was characterized by a component of depression was measured by the Snaith-Hamilton Pleasure Scale (SHAPS).The SHAPS questionnaire is composed of 14 questions, the total score of the SHAPS varies between 0 and 14. Severe anhedonia will be observed if the SHAPS score is strictly greater than 5.

SECONDARY OUTCOMES:
Evolution of the subject's mood | 84 days
  Evolution of the mood of subjects measured by the Brief Mood Introspection Scale (BMIS).Each "positive" item (Dynamic, Happy, Compassionate, Content, Energetic, Quiet, Affectionate and Vivid) is rated from 1 "Not at all" to 4 "Absolutely". Each item "negative" (Sad, Tired, Melancholic, Excited, Exhausted, Grumpy, Nervous and Annoyed) is inversely rated from 1 "quite" to 4 "not at all". The BMIS questionnaire is composed of 16 questions, and will be calculated by adding the answers of these 16 items. The BMIS score varies between 16 and 64.
The effect on work and other activities | 84 days
  The effect on work and other activities according to item 7 of the Hamilton Rating Scale for Depression (HAM-D).The HAM-D is a scale for depression composed of 17 questions and varies between 0 and 58.
  The HAM-D score will also be classified into 5 classes according to the following model:
  0-7 None; 8-13 Light; 14-18 Moderate; 19-22 Severe; > 23 Very severe
Evolution of the components of depression | 84 days
  Evolution of the components of depression is measured by the Quick Inventory of Depressive Symptomatology -Self-Report (QIDS-SR).QIDS-SR questionnaire is composed of 16 questions. Each answer is scored from 0 to 3. The symptomatology is more important with a higher score. The total score fluctuates between 0 and 27.
  The QIDS score will also be classified into 5 classes according to the following model:
  0-5 None; 6-10 Lightweight; 11-15 Moderate; 16-20 Severe; > 20 Very severe
Evaluation of subject's satisfaction | 84 days
  Subject's satisfaction with the treatment was evaluated by the Patient Global Improvement Impression (PGII)
Evaluation of product's tolerance | 84 days
  The evaluation of product's tolerance for the whole period of the trial is done by the reporting of Serious Adverse Event if any
Evaluation of the investigator's opinion | 84 days
  Evaluation of the investigator's opinion is measured by the Clinical Global Improvement Impression (CGII)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allaert FA, Demais H, Collen PN. A randomized controlled double-blind clinical trial comparing versus placebo the effect of an edible algal extract (Ulva Lactuca) on the component of depression in healthy volunteers with anhedonia. BMC Psychiatry. 2018 Jun 28;18(1):215. doi: 10.1186/s12888-018-1784-x. PMID 29954354